CLINICAL TRIAL: NCT01112657
Title: A Prospective, Observational Study On The Progression Of Clinically Isolated Syndrome (CIS) To Multiple Sclerosis Over A 2-year Period
Brief Title: An Observational Study on the Progression of Clinically Isolated Syndrome to Multiple Sclerosis Over a 2-year Period
Acronym: NEO
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200077-504
Record Dates: First submitted 2010-03-10; First posted 2010-04-28 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Clinical isolated syndrome; Demyelination
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, multicentric, observational study with a 2 years recruitment period. The purpose of the study is to observe the multiple sclerosis (MS) progression of subjects since their first episode of neurological event and secondly, to determine status of anti-AQP4 immunoglobulin (IgG) antibody in MS subjects.

DETAILED DESCRIPTION:
Multiple sclerosis is chronic, inflammatory disease of the central nervous system (CNS) characterised by areas of demyelination, or plaques, in the CNS. In 85% of subjects who later develop MS, clinical onset is with an acute or subacute episode of neurological disturbance due to a single white-matter lesion (e.g. optic neuritis, or an isolated brainstem or partial spinal-cord syndrome). This presentation is known as a Clinically Isolated Syndrome (CIS). Because a CIS is typically the earliest clinical expression of MS, research on subjects with a CIS may provide new insights into early pathological changes and pathogenetic mechanisms that might affect the course of the disorder.

In the group of subjects with optic-spinal MS (OSMS), the main lesions are typically confined to the optic nerve and spinal cord. In Asians, OSMS has similar features to the relapsing remitting form of neuromyelitis optica (NMO) seen in Westerners. It is still a matter of debate whether NMO represents a disease entity in itself or whether it is a subform of MS. Early differentiation of NMO from MS is highly desirable, as treatment options and prognoses differ widely. Recently, a new serum autoantibody (NMO-IgG) has been detected in NMO subjects. The binding sites of this autoantibody were reported to colocalize with aquaporin 4 (AQP4) water channels. Optic-spinal MS is sometime suggested to be NMO based on the frequent detection of the anti-AQP4 IgG antibody. In Taiwan, study has shown that 56% of MS subjects were of the optic-spinal type.

OBJECTIVES

The study is designed firstly, to observe the MS progression of subjects since their first episode of neurological event and secondly, to determine status of anti-AQP4 IgG antibody in MS subjects.

Primary objective:

* To describe the progression of subjects who have experienced a CIS to MS over a 2-year period

Secondary objectives:

* To assess the relationship between CIS and MS including optic-spinal MS (OSMS)
* To determine the status of anti-AQP4 IgG antibody in subjects who convert to MS

Each subject shall be followed up for 2 years after enrolment. At baseline, routine examinations shall be performed to confirm subject's neurological episode. After the baseline visit, the subject shall be instructed to return for further examination if he/she experiences a relapse. During the follow-up examinations, the treating physician shall determine whether the subject fulfil the diagnostic criteria for MS.

If subject is being diagnosed with MS, he/she shall be considered as reaching the end of his/her study participation. Further management of the MS condition will be at the discretion of the treating physician. During 2-year follow-up period, telephone calls to the subject shall be made quarterly to assess subject's neurological and/or visual status and to remind subject that he/she need to return for evaluation in the event of a relapse. All data will be collected using a standardised case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 6-60 years, both inclusive
* Subjects who have experienced a single, first clinical event potentially suggestive of MS within the last 2 years from study entry. The event must be a new neurological abnormality present for at least 24 hours, either mono- or polysymptomatic, other than paresthesia or vegetative dysfunction
* Subjects who have given written informed consent.

Exclusion Criteria:

* Subjects with the diagnosis of MS
* Subjects with other disease that could better explain the subject's signs and symptoms
* Subjects who are scheduled to participate in any interventional treatment trial
* Subjects who have any condition that could interfere with MRI evaluation

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who have experienced a single, first clinical event potentially suggestive of MS within the last 2 years from study entry.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2008-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who convert to multiple sclerosis (MS), defined by McDonald criteria (Version 2005), over 2 years from the first episode of Clinically Isolated Syndrome (CIS) | Baseline to 2 years
  At each and every visit, routine neurological and or ophthalmologic examinations will be performed to determine whether subject has progress to MS.

SECONDARY OUTCOMES:
Duration between first episode of neurological event and diagnosis of MS | Baseline to 2 years
Proportion of subjects with conventional MS and optic-spinal MS (OSMS) | Baseline to 2 years
Proportion of subjects with anti-AQP4 IgG antibody | Baseline to 2 years
  Blood samples shall be taken at baseline, 12-16 weeks after baseline and end of study (for subjects who converted to MS) for anti-AQP4 IgG antibody measurements
Association between baseline demographics/disease characteristics and progression to MS | Baseline to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Piao Tsai, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (6):
- Taiwan (6):
  - Kaohsiung Medical University, Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang-Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital - Linkou Branch, Taoyuan District